CLINICAL TRIAL: NCT05382221
Title: Breathe 2 Project 3: Comprehensive Chronic Care
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Wisconsin, Madison (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2022-0124; Protocol Version 10/12/2023 (Other: UW Madison); A534253 (Other: UW Madison); 2P01CA180945-06 (NIH)
Record Dates: First submitted 2022-05-16; First posted 2022-05-19 (Actual); Last update posted 2025-12-18 (Actual); Status verified 2025-12

CONDITIONS: Smoking Cessation; Smoking Abstinence
Keywords: Chronic Care Tobacco Treatment; Standard of Care; Reduction Treatment; Motivation Phase Treatment
MeSH Terms: conditions — Smoking Cessation | interventions — Standard of Care

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Comprehensive Chronic Care (Experimental): ongoing proactive outreach designed to provide support and information about evidence-based smoking treatment, with access to individually validated treatments that are appropriate for patients who are: 1) unwilling quit but willing to reduce; 2) ready to quit; and 3) recovering from an unsuccessful quit attempt
  Interventions: Other: Comprehensive Chronic Care
- Standard Care (Active Comparator): involves one offer of cessation treatment (8 weeks of nicotine patch plus referral to the tobacco quit line), annually
  Interventions: Other: Standard Care

INTERVENTIONS:
Other: Comprehensive Chronic Care — Those randomized to CCC will receive smoking treatment offers via the following routes: 1) Four Outreach Calls from a Health Counselor at 4, 8, 12, and 14 months post-study enrollment; 2) Four texts and/or mailings (depending on healthcare system preferences) over 14 months. These outreach contacts will offer cessation treatment or reduction treatment.
  Arms: Comprehensive Chronic Care
Other: Standard Care — one offer of cessation treatment annually
  Arms: Standard Care

SUMMARY:
This study will evaluate Comprehensive Chronic Care (CCC), a healthcare treatment approach designed to increase smoking treatment engagement and abstinence among primary care patients who smoke. This research will compare CCC with Standard of Care (SC) on the following outcomes: abstinence at 18 months (primary outcome), treatment reach, and cost-effectiveness. Participation in the study will last 18 months.

DETAILED DESCRIPTION:
This project is a 2-arm randomized controlled trial (RCT) designed to evaluate whether Comprehensive Chronic Care (CCC), relative to Standard Care (SC), increases smoking abstinence and treatment use in primary care patients who smoke. The aims are as follows:

* Primary Aim

  * Aim 1: To determine whether Comprehensive Chronic Care (CCC), relative to Standard Care (SC), significantly improves biochemically confirmed 7-day point-prevalence smoking abstinence at 18 months post-enrollment.
* Secondary Aims

  * Aim 2: To determine the effects of CCC relative to SC on: cost-effectiveness and 7-day point-prevalence smoking abstinence at 6- and 12-months (biochemically confirmed) post-enrollment.
  * Aim 3: To compare CCC with SC on cessation treatment use over 18 months of treatment access.

Comprehensive Chronic Care (CCC) provides ongoing proactive outreach designed to provide support and information about evidence-based smoking treatment, with access to individually validated treatments that are appropriate for patients who are: 1) unwilling quit but willing to reduce; 2) ready to quit; and 3) recovering from an unsuccessful quit attempt.

Standard Care (SC) involves one offer of cessation treatment per year (8 weeks of nicotine patch plus referral to the tobacco quit line).

ELIGIBILITY:
Inclusion Criteria:

* On smoking registry at a participating clinic OR report current smoking at a clinic visit
* Smoked cigarettes every day in the past 30 days (with or without other forms of tobacco or nicotine)
* Able to participate in informed consent activities (e.g., reports understanding the nature of the study and consent)
* Able to speak and read English.

Exclusion Criteria:

* Activated healthcare power of attorney or cognitive impairment that would preclude informed consent.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 979 (Actual)
Dates: Start 2022-08-08 (Actual); Primary Completion 2025-09-25 (Actual); Study Completion 2025-09-25 (Actual)

PRIMARY OUTCOMES:
Number of Participants with biochemically confirmed point-prevalence abstinence at 18 months | up to 18 months
  Group differences in abstinence at 18 months will be evaluated using logistic regression.

SECONDARY OUTCOMES:
Number of Participants with 7-day point-prevalence abstinence at 6 months | 6 months
  At 6 months, participants will be asked whether they have smoked in the past 7 days
Number of Participants with 7-day point-prevalence abstinence at 12 months | 12 months
  At 12 months, participants will be asked whether they have smoked in the past 7 days
Group differences in Cessation Treatment | Up to 18 months
  Group differences in cessation treatment use will be evaluated using logistic regression analysis. Initiating greater than 0 Cessation calls will be coded as binary (use vs. no use).
Total Cost of Intervention | Up to 18 months
  Incremental resource costs related to the CCC intervention include Health Counselor/staff time, administration, staff training, recruitment, and medication. Methods recommended by the United States Panel on Cost-Effectiveness in Health and Medicine will be utilized. Costs will be measured from a societal perspective using direct observational data of health system resource use. Cost estimates will be converted to a common year.
Cost Effectiveness measured by incremental cost-effectiveness ratio (ICER) | Up to 18 months
  Cost per additional person who quits smoking, for the CCC vs. SC. The ICER is calculated as the difference in total costs between CCC and SC divided by the difference in 18-month quit rates.

CONTACTS AND LOCATIONS:
Overall Officials: Jessica Cook, PhD, Principal Investigator — UW Center of Tobacco Research and Intervention
Locations (2):
- United States (2):
  - UW Health, Madison, Wisconsin
  - Advocate Aurora, Milwaukee, Wisconsin

IPD SHARING:
Plan to Share IPD: No

DOCUMENTS (1):
  • Informed Consent Form (2023-07-28): https://cdn.clinicaltrials.gov/large-docs/21/NCT05382221/ICF_000.pdf